CLINICAL TRIAL: NCT04222023
Title: Intravenous Immunoglobulins for Prevention of BKV Infection in Kidney Transplant Recipients According to BKV Genotype-specific Neutralizing Antibody Titers at the Day of Transplantation: A Multicenter Study
Brief Title: Intravenous Immunoglobulins for Prevention of BKV Infection in Kidney Transplant Recipients According to BKV Genotype-specific Neutralizing Antibody Titers at the Day of Transplantation.
Acronym: BKANIG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6997
Record Dates: First submitted 2019-12-19; First posted 2020-01-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVIG group (Experimental): Administration of a single dose of IVIG at day 10+/- 4 days, day 41 +/- 7 days and day 62 +/- 7 days. The dose of IVIG is defined according the donor BKV genotype: genotype I: 0.4 g/Kg/day; genotype II and IV: 1g/kg/day.
  Interventions: Drug: Intravenous immunoglobulins (IVIG)
- Control group (No Intervention)

INTERVENTIONS:
Drug: Intravenous immunoglobulins (IVIG) — Experimental group: administration of a single dose of IVIG at:
  * Day 10+/- 4 days
  * Day 41 +/- 7 days
  * Day 62 +/- 7 days The dose of IVIG is defined according the donor BKV genotype: genotype I: 0.4 g/Kg/day; genotype II and IV: 1g/kg/day.
  Arms: IVIG group

SUMMARY:
BK virus-associated nephropathy (BKVAN), a consequence of the strong immunosuppressive therapy given after kidney transplantation (KT), represents a growing medical problem in the KT setting. BKV replication occurs in 30-50% of recipients with progression to BKVAN in up to 10% of patients which ultimately leads to graft dysfunction and loss. Furthermore, early BKV replication after transplantation increases the risk of late acute rejection. At present, there are no BKV-specific antiviral therapies available. The current management of BKVAN relies on preemptive adaptation of immunosuppression according to viral load monitoring. However, due to its delayed nature, this empirical strategy is not always successful, and can increase the risk of donor specific antibodies, graft rejection and death. In a prospective longitudinal study, the investigators have demonstrated that the amount and kinetics of BKV genotype-specific neutralizing antibody (NAb) titers influence BKV disease severity after KT; and defined a cutoff NAb titer value of 4 log10 that allows stratification of recipients into lower and higher BKV disease risk groups prior to KT. Furthermore, our data on donor/recipient pairs provide support for the view reported by recent studies that early BKV replication in kidney transplant recipients is of donor origin. These data support the potential benefit of administering NAbs as a preventive strategy against BKV infection. The investigators and others have demonstrated the presence of high titers of BKV NAbs in commercial intravenous immunoglobulins (IVIG). The investigators further evaluated the titer of BKV NAbs in plasma samples of transplant recipients after administration of IVIG. The investigators demonstrated that all patients show an increase of NAb titers in plasma after IVIG administration. The aim of the investigators study is to investigate the efficacy of IVIG for prevention of BKV viremia after KT according to pre-transplant BKV genotype-specific NAb titers against the donor's BKV strain. The study is a multicentric prospective randomized open trial evaluating the impact of administration of IVIG for prevention of BKV viremia compared to no specific treatment in kidney transplant recipients harboring neutralizing antibody titers (NAbs) ≤ 4log10 against the BKV donor's genotype. Recipients harboring BKV NAb titer ≤ 4log10 against the BKV genotype of their matched donor and negative or non-detectable BKV load in blood at day of transplantation will be randomized to receive (experimental group) or not (control group) IVIG treatment. In the experimental group, patients will receive a single dose of IVIG at day 10+/- 4 days, day 41 +/- 7 days and day 62 +/- 7 days. The dose of IVIG is defined according the donor BKV genotype: genotype I: 0.4 g/Kg/day; genotype II and IV: 1g/kg/day.

The incidence of BKV viremia (> 4 log10 copies/mL) 6 months after transplantation will be evaluated and compared between the two groups.

ELIGIBILITY:
Inclusion criteria:

* Adult patients (> 18 years)
* Kidney transplant recipients, including multiple organ transplant patients
* Patients able to understand the purpose and the risks of the study, fully informed and having written informed consent
* Negative pregnancy test
* Affiliated to a medical insurance scheme

Exclusion criteria:

* BKV nephropathy during a previous transplantation in the past 5 years
* HLA and ABO-incompatible kidney transplant recipients undergoing desensitization with rituximab and/or plasmapheresis before transplantation or susceptible to receive such therapy after transplantation
* Patients with high risk of post- transplant Focal Segmental glomerulosclerosis recurrence
* Patient with hyperprolinemia
* Allergy or known intolerance to IVIG
* Pregnant or breast feeding women
* Adults under guardianship or limited guardianship
* Currently participating in another clinical trial investigating drugs (observational studies are not considered as an exclusion criterion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2022-08-21 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
The incidence of BKV viremia | BKV viremia will be measured at the day of transplantation at day 10
The incidence of BKV viremia | BKV viremia will be measured at the day of transplantation at day 41
The incidence of BKV viremia | BKV viremia will be measured at the day of transplantation at day 62
The incidence of BKV viremia | KV viremia will be measured at the day of transplantation at months 3
The incidence of BKV viremia | BKV viremia will be measured at the day of transplantation at months 6
The incidence of BKV viremia | BKV viremia will be measured at the day of transplantation at months 12

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Helle F, Aubry A, Morel V, Descamps V, Demey B, Brochot E. Neutralizing Antibodies Targeting BK Polyomavirus: Clinical Importance and Therapeutic Potential for Kidney Transplant Recipients. J Am Soc Nephrol. 2024 Oct 1;35(10):1425-1433. doi: 10.1681/ASN.0000000000000457. Epub 2024 Jul 9. PMID 39352862